CLINICAL TRIAL: NCT03329040
Title: Is Primiparity a Risk Factor for Neonatal Hyperbilirubinemia?
Status: Completed | Type: Observational
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Principal Investigator, Erez Nadir, MD, Neonatologist, Hillel Yaffe Medical Center
Other Study IDs: 0090-17-HYMC-CTIL
Record Dates: First submitted 2017-10-30; First posted 2017-11-01 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Hyperbilirubinemia, Neonatal
Keywords: Hyperbilirubinemia; Primiparity; multiparity
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal; Hyperbilirubinemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primipara mothers: Infant to primipara mothers, i.e. the first infant to the mother - No intervention
  Interventions: Other: No Intervention.
- Multipara mothers: Infant to multipara mothers, i.e. not the first infant to the mother - No intervention
  Interventions: Other: No Intervention.

INTERVENTIONS:
Other: No Intervention. — No intervention.

SUMMARY:
Neonatal hyperbilirubinemia elongates hospital stay and may require treatment. The investigators noticed that bilirubin levels were higher among infants of primipara mothers than among multipara mothers. As this data is dichotomic and easy to produce, and may influence the maintenance, the investigators decided to find out if primiparity is a risk factor for neonatal hyperbilirubinemia. The investigators intend to collect data from patient files during one year, and compare the bilirubin levels and length of stay between newborns to primipara mothers and multipara mothers.

DETAILED DESCRIPTION:
Neonatal hyperbilirubinemia elongates hospital stay and may require treatment. The investigators noticed that bilirubin levels were higher among infants of primipara mothers than among multipara mothers. As this data is dichotomic and easy to produce, and may influence the maintenance, the investigators decided to find out if primiparity is a risk factor for neonatal hyperbilirubinemia. The investigators intend to collect data from patient files during one year, and compare the bilirubin levels and length of stay between newborns to primipara mothers and multipara mothers.

ELIGIBILITY:
Inclusion Criteria:

* All infants that were born during one year in a single medical center and were transferred to well baby nursery, and were discharged from the well baby nursery.

Exclusion Criteria:

* Infants who were transferred to neonatal intensive care unit due to any reason.
* Infants whose mother could not take care of them (due to admission to intensive care unit, or due to adoption)

Max Age: 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants who were born during one year, in a single medical center
Sampling Method: Non-Probability Sample
Enrollment: 4369 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
Length of stay of the infant | 2 weeks
  Length of stay of the infant

SECONDARY OUTCOMES:
Highest bilirubin level | 2 weeks
  Highest bilirubin level
Age at highest bilirubin level | 2 weeks
  Age at highest bilirubin level

CONTACTS AND LOCATIONS:
Overall Officials: Erez Nadir, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe medical center, Hadera, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No
Unidentified data will be collected in an Excel workbook

REFERENCES:
- [Background] Amos RC, Jacob H, Leith W. Jaundice in newborn babies under 28 days: NICE guideline 2016 (CG98). Arch Dis Child Educ Pract Ed. 2017 Aug;102(4):207-209. doi: 10.1136/archdischild-2016-311556. Epub 2017 Feb 8. No abstract available. PMID 28179382
- [Background] Brotman DJ, Walker E, Lauer MS, O'Brien RG. In search of fewer independent risk factors. Arch Intern Med. 2005 Jan 24;165(2):138-45. doi: 10.1001/archinte.165.2.138. PMID 15668358
- [Background] American Academy of Pediatrics Subcommittee on Hyperbilirubinemia. Management of hyperbilirubinemia in the newborn infant 35 or more weeks of gestation. Pediatrics. 2004 Jul;114(1):297-316. doi: 10.1542/peds.114.1.297. PMID 15231951